CLINICAL TRIAL: NCT07200973
Title: People & Place: Impacts on Substance Use and HIV Outcomes in Los Angeles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Pamina Mae Gorbach, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA061345 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: HIV

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted LINK-LA Peer Case Management (Experimental): LINK-LA Peer Case Management Intervention, adapted for people living with HIV who use substances
  Interventions: Behavioral: Adapted LINK LA Peer Navigator

INTERVENTIONS:
Behavioral: Adapted LINK LA Peer Navigator — Our study will adapt the LINK LA peer navigation intervention (NCT01406626) for the current context (e.g., HIV care provision, substance use risk environments, etc.) and measure its effects on participants' HIV and substance care engagement.

SUMMARY:
This study will implement an adapted peer navigation intervention to improve linkage to and retention in HIV care for people living with HIV who experience substance use within Los Angeles County.

DETAILED DESCRIPTION:
People living with HIV often experience additional challenges when substance use is also part of their lives. Staying in consistent HIV care is essential for maintaining health, but this can be complicated when services are difficult to access or require navigating multiple systems. In a large, urban county like Los Angeles, where clinics and treatment centers are widely dispersed, people may need to travel long distances, rely on limited transportation, or attend separate locations for HIV care and substance use treatment. These factors can create real barriers to staying engaged in care, even when services are technically available. The "People & Place" study is designed to better understand how individuals living with HIV move through Los Angeles to obtain their care, and how the organization of healthcare services and policies influence those experiences. The study examines the role and impact of peer case managers-individuals with relevant, compatible experiences who can guide and support participants as they navigate the healthcare system. Peer case managers may be able to reduce barriers by helping patients find care within their nearby communities, strengthening connections with providers, and encouraging continuity of treatment.

The project represents a collaboration between researchers at University of California, Los Angeles (UCLA), the University of California, Santa Barbara (UCSB), and a local HIV clinic, bringing together expertise in medicine, public health, and community-based care. By combining academic research with input from patients and healthcare providers, this research aims to create practical and effective strategies for reducing barriers such as distance, transportation, and fragmented services, ultimately improving the accessibility, coordination and patient-centeredness of healthcare delivery for people living with HIV who also use substances.

Specific Aims include:

Aim 1. Connect existing policies and conditions (e.g., heat exposure, policing, and economic distribution) with geospatial patterns of health outcomes among people living with HIV via compilation of secondary data with new data collected among people living with HIV through an innovative "activity space" survey. These harmonized data will document spatial associations between local, state, and federal policies and contemporary contextual determinants of health at the neighborhood level and identify how perceptions of territorial reputations, and local spaces influence preferences for HIV care and SU harm reduction services.

Aim 2. Qualitatively assess the HIV and substance use care experience among people living with HIV (n=30) as well as staff members at a large HIV care clinic in LA (n=15) via qualitative interviews (N=45 total) to examine how experiences and perceptions of space influence service use and movement through HIV and substance use hotspots, in other words: the geography of care.

Aim 3. Adapt and pilot the evidenced based intervention, LINK LA (NCT01406626), to examine the role of a compatible peer case management intervention on HIV and substance use outcomes. Activities of this aim include: (a) undertaking a process of intervention adaptation utilizing results from qualitative interviews in Aim 2 with clinic staff and people living with HIV, and conduct theatre testing of the intervention, (b) piloting the adapted intervention among N=250 people living with HIV to assess acceptability and feasibility and assess the preliminary impacts of the adapted intervention on HIV and substance use outcomes, and (c) examining the relationship between the distance of where participants live and their choice of an enhanced HIV and substance use care experience based on an adapted intervention. Results will identify patterns in HIV and substance use care choices and outcomes across LAC's geographically broad neighborhoods and determine if an intervention can modify such choices and outcomes. The intervention is hypothesized to result in greater linkage to care, increased self-reported ART adherence, and decreased levels of HIV RNA viral load in comparison to pre-intervention periods.

ELIGIBILITY:
Inclusion Criteria:

* Living with HIV
* Assigned male sex at birth
* Willing to return for follow-up study visits every six months as long as the study is ongoing and be available to return for all study visits, barring unforeseen circumstances
* Willing and able to provide written informed consent to take part in the study
* Willing and able to provide adequate information for locator purposes
* Willing to undergo repeat HIV viral load testing at select study visits
* Willing to undergo substance use testing at each study visit

Exclusion Criteria:

* Born biologically female
* Unwilling or unable to provide reliable contact information
* Unwilling to provide urine or blood
* Any other condition or prior therapy that, in the opinion of the research staff would preclude informed consent, make study participation unsafe, make the individual unsuitable for the study or unable to comply with the study requirements. Such conditions may include, but are not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, or cerebral disease, among others

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with HIV Viral Suppression | From enrollment to the end of intervention period at 24 weeks
  Measured via HIV Viral Load (copies/mL)
Number of Participants with HIV Care Adherence | From enrollment to the end of intervention period at 24 weeks
  Participants' engagement in their HIV care, defined by attendance at scheduled HIV medical appointments

SECONDARY OUTCOMES:
Number of Participants with HIV Antiretroviral (ART) Adherence | From enrollment to the end of intervention period at 24 weeks
  Participants self-reported adherence to daily ART medication within the past 7 days
Number of Participants with Recent Substance Use | From enrollment to the end of intervention period at 24 weeks
  Results of rapid urine toxicology testing conducted at scheduled study visits